CLINICAL TRIAL: NCT01201616
Title: The Effects of a High Fat, Low Carbohydrate or a Low Fat, High Carbohydrate Diet on Mood Cognition and Appetite
Brief Title: The Effects of Diet on Mood, Cognition and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Mars, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RIS030426a
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognitive function; mood; women; high fat diet; high carbohydrate diet
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat, low carbohydrate diet (Experimental): Fats intake 55% , Protein 17% and carbohydrate 28% of total energy
  Interventions: Other: High Fat Low Carbohydrate Diet
- Low fat, high carbohydrate diet (Active Comparator): Fat intake 20%, Protein 17% and carbohydrate 63% of total energy intake
  Interventions: Other: Low fat High Carbohydrate Diet

INTERVENTIONS:
Other: High Fat Low Carbohydrate Diet — 55% total energy intake from fats, 17% from protein and 28% from carbohydrate
  Other Names: HFLC Diet
  Arms: High fat, low carbohydrate diet
Other: Low fat High Carbohydrate Diet — 20% total energy intake from dietary fats, 17% from protein and 63% from carbohydrate
  Other Names: LFHC Diet
  Arms: Low fat, high carbohydrate diet

SUMMARY:
A previous study has found that the consumption of a high fat, low carbohydrate meal results in increased feelings of calmness, friendliness and an increase in subjective energy levels in comparison to a low fat, high carbohydrate meal. The purpose of this study is to investigate whether a high fat, low carbohydrate diet for a longer duration (of 2 weeks) can enhance or sustain these changes in comparison to a low fat, high carbohydrate meal.

DETAILED DESCRIPTION:
Research has shown that consuming breakfasts high in either fat or carbohydrates can affect a persons memory, mood and ability to concentrate (Benton & Parker, 1998, Politt & Mathews, 1998). Our previous study investigating the effect of a high fat, low carbohydrate (HFLC) meal in comparison to a low fat, high carbohydrate (LFHC) meal found that the HFLC meal resulted in significantly increased feelings of calmness, friendliness and a reduction in feelings of anger, and an increase in subjective energy levels in comparison to a LFHC meal. However, the chronic effects of a HFLC or LFHC diet has not been studied. This purpose of this study is to investigate whether a 2 week diet high in either fat or carbohydrates improves cognition/memory and mood. It is hypothesised that the prolonged feeding of a HFLC diet will attenuate the response seen after a HFLC meal was provided.

Twenty healthy women are required to attend the School of Biomedical Sciences on seven occasions.

The first visit will involve screening tests for suitability for inclusion in the study and written, informed consent will be obtained. Weight, height and blood pressure will be measured and a 5ml blood sample will be collected for full blood count, urea, electrolytes and random blood glucose assessment. Subjects will be asked to complete questionnaires regarding general health, eating habits, mood and medical history. Following the screening visit, subjects will be asked to record their habitual food intake and physical activity pattern for a 3 day period (2 weekdays and 1 weekend day. They will then attend the laboratory on 6 further occasions, once for a familiarisation visit and for the 5 study visits.

The familiarisation visit is required to ensure that subjects are comfortable and familiar with using the cognitive tests which will be administered.

Subjects will be provided with a menu of foods to consume as their evening meal prior to study visits, based on 30% total energy expenditure. This meal will be based on foods the subject recorded in the completed food diary and will contain approximately 15% of total energy from protein, 55% from carbohydrate and 30% from fat. Before study visits subjects will be instructed to consume this standardised meal as their last meal of the day before 20.00 on the previous evening. After they have consumed this meal they are instructed not to consume any foods or drinks apart from water until they arrive at the lab.

Subjects will arrive (fasted) at the lab at 08.00 on the morning of each study visit. A cannula will be inserted retrograde into a hand vein, after prior infiltration at insertion site with 1% lidocaine. The hand will be placed in a heated box, and remain there throughout the trial, to obtain arterialised venous blood samples. The cannula will be kept patent with a slow infusion of 0.9% saline, and samples will be taken via a three-way tap.

Subjects will then be either given a HFLC, or a LFHC breakfast, the order being randomised. The HFLC breakfast will be provided on study days before and after the HFLC diet intervention, and the LFHC breakfast will be provided on study days before and after the LFHC diet intervention.

Water will be freely available throughout the day. Every 30 minutes subjects will be asked to complete a set of visual analogue scales designed to assess subjective mood and satiety, a 15ml blood sample will be taken for the measurement of glucose, insulin, ghrelin, free fatty acids, glucagon, cholecystokinin (CCK), Glucagon-like peptide 1 (GLP-1), cortisol, adrenaline and noradrenaline. A 3ml sample will be taken every 15minutes for the first 90 minutes, for the analysis of insulin and glucose. A baseline sample for triglycerides and cholesterol will be taken at the beginning of each study visit. Cognitive tests (measuring attention reaction times and vigilance) will be completed 0, 45, 90 and 135 minutes minutes after the provision of breakfast. After 180 minutes, the cannula will be removed and subjects will be free to leave the lab.

Subjects will be provided with either a HFLC diet or a LFHC diet to consume for 2 weeks. These diets will be designed to meet subjects energy requirements. After consuming the diet for 2 weeks (diets will comprise of 3 meals and 3 snacks per day), subjects will return to the laboratory for the second study visit. Subjects will be provided with a set of visual analogue scales to complete on days 4, 8 and 12 of the intervention period. Subjects will then return to their habitual diets for 2 weeks, before completing the second intervention.

Subjects will also be asked to come to the laboratory for an additional study visit either 2 days before visit 1 or two days before visit 3, where they will be consume their habitual breakfast instead of a HFLC or LFHC breakfast.

During both the 2 week intervention periods, subjects will be asked to consume only the food provided, no other drinks, including alcohol and caffeinated drinks, may be consumed. If subjects are habitual tea/coffee drinkers then they may consume a maximum of 3 cups of tea/coffee a day (unsweetened, with milk from their daily allocation) and be asked to maintain this over both arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* female
* BMI 18.5-25kg/m2
* aged 18-45 years
* regular breakfast eaters
* regular menstrual cycle
* healthy

Exclusion Criteria:

* Significant gastrointestinal disease, gastrointestinal surgery, diabetes or any other significant major medical morbidity
* History of significant eating disorder (anorexia, bulimia)
* Habitual dietary protein intake >20% of total energy intake
* pregnancy or breast feeding
* anaemia (Hb <11.5g/dL)
* random blood glucose concentration >8mmol/l
* no medication use other than contraception
* significant weight loss/gain (>14lb in previous 3 months)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Clear-headedness | after 2 week intervention period
  Subjective mood measurement, assessed using visual analogue scale, in response to a test meal

SECONDARY OUTCOMES:
Reaction time | after 2 week intervention
  cognitive function measurement, assessed using choice reaction time, in response to a test meal

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Notts, United Kingdom

REFERENCES:
- [Background] Benton D, Parker PY. Breakfast, blood glucose, and cognition. Am J Clin Nutr. 1998 Apr;67(4):772S-778S. doi: 10.1093/ajcn/67.4.772S. PMID 9537627
- [Background] Pollitt E, Mathews R. Breakfast and cognition: an integrative summary. Am J Clin Nutr. 1998 Apr;67(4):804S-813S. doi: 10.1093/ajcn/67.4.804S. PMID 9537633